CLINICAL TRIAL: NCT02029027
Title: Evaluation de l'intérêt de l'électrostimulation Intra-vaginale à Domicile Par Rapport à Une Prise en Charge Habituelle Dans la Prise en Charge de Patientes Incontinentes Ayant bénéficié d'Une rééducation périnéale
Brief Title: Interest of Intravaginal Electro-stimulation at Home by GYNEFFIK® Compared to Usual Care in Incontinent Patients With Prior Perineal Reeducation
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Effik (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2012-A00235-38
Record Dates: First submitted 2014-01-06; First posted 2014-01-07 (Estimated); Last update posted 2014-01-07 (Estimated); Status verified 2014-01

CONDITIONS: Urinary Stress Incontinence; Urinary Mixed Incontinence
Keywords: Urinary Stress Incontinence; Urinary Mixed Incontinence
MeSH Terms: conditions — Urinary Incontinence, Stress

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- GYNEFFIK(R) (Experimental): 30 min-session of vaginal electro-stimulation by GYNEFFIK thrice a week for 6 months (except during menstrual periods)
  Interventions: Device: GYNEFFIK(R)
- Usual Care (Other): Any treatment / physiotherapy sessions / muscular training ... usually recommended and/or prescribed by the patient's general practitioner or gynaecologist with the exception of vaginal electro-stimulation
  Interventions: Other: Usual Care

INTERVENTIONS:
Device: GYNEFFIK(R) — Vaginal electro-stimulation medical device
  Arms: GYNEFFIK(R)
Other: Usual Care — Any treatment / physiotherapy sessions / muscular training ... usually recommended and/or prescribed by the patient's general practitioner or gynaecologist with the exception of vaginal electro-stimulation
  Arms: Usual Care

SUMMARY:
The aim of this study is to assess the benefit of GYNEFFIK®, a perineal electro-stimulator, during this home-care phase. Women with stress urinary incontinence (UI) or with mixed UI (composed predominantly of stress UI), that responded to physiotherapy were included in this study in two parallel groups. The groups followed a self-reeducation program, with or without GYNEFFIK® electro-stimulation sessions. The comparison of the two groups was based on the rate of women for whom the benefit of the initial perineal reeducation was maintained.

ELIGIBILITY:
Inclusion Criteria:

* out-patient over 18 years old, having understood and signed the Informed Consent Form
* seen for urinary stress incontinence or urinary mixed incontinence (with a major stress incontinence part) troubles
* spontaneously asking for help
* who can be followed for a long time

Exclusion Criteria:

* Urinary Incontinence (UI) found out during medical interviewing without spontaneous complaint
* Urinary troubles due to neurological pathology (stroke, multiple sclerosis, ...)
* UI due to congenital malformation
* UI having led to surgery
* UI treated in the last 6 months
* UI within 24 weeks of Past Partum
* Pelvic surgery within 12 months
* On-going inflammatory or infectious neoplastic disease
* Perineal hypoesthesia
* Local conditions prohibiting the use of an intra-vaginal device (vaginal atrophia, continuous metrorrhagia, vaginal prolapse > 2°, ...)
* Pacemaker use
* Women of child bearing potential without effective method of contraception or planning to get pregnant in the next 12 months
* Intravaginal contraception
* Mental impairment or inability to understand or follow study instructions
* Patient who may not come back to the study visits
* Patient already enrolled for another study or having been enrolled in another clinical study in the past 3 months

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 163 (Actual)
Dates: Start 2012-08; Primary Completion 2014-02 (Estimated); Study Completion 2014-02 (Estimated)

PRIMARY OUTCOMES:
Non-Worsening of ICIQ + Ditrovie Scales' Scores | 6 Months (or last measurement if premature ending)
  The primary outcome is defined as the non worsening of the ICIQ (International Consultation on Incontinence modular Questionnaire) scale's score AND the DITROVIE scale's score (a specific scale to evaluate the perturbation of the quality of life during urinary troubles).
  The scores will be considered as maintained if they didn't increase more than 10% with the following calculation:
  ICIQ variation (%) = 100 x (ICIQ_M6 - ICIQ_D0)/ICIQ_D0
  DITROVIE variation (%) = 100 x (DITROVIE_M6 - DITROVIE_D0)/(DITROVIE_D0 -10)

SECONDARY OUTCOMES:
ICIQ Score | 6 Months (or last measurement if premature ending)
  Quantitative analyses:
  * difference = ICIQ_M6 - ICIQ_D0
  * variation (%)= 100 x (ICIQ_M6 - ICIQ_D0)/ICIQ_D0
  Qualitative analysis
  * % of patients with a variation % <-10%, between -10% and +10%, >10%
DITROVIE Score | 6 Months (or least measurement if premature ending)
  Quantitative analyses:
  * difference = DITROVIE_M6 - DITROVIE_D0
  * variation (%)= 100 x (DITROVIE_M6 - DITROVIE_D0)/(DITROVIE_D0 - 10)
  Qualitative analysis
  * % of patients with a variation % <-10%, between -10% and +10%, >10%
ICG score | 6 Months (or last measurement if premature ending)
  The ICG (clinical global impression) score is the subjective impression of the patient regarding the evolution of her own clinical condition. It will be determined between inclusion and M6 (or the last visit).
SF-12 Health Survey (Medical Outcomes Study Short-Form General Health Survey) | 6 Months (or last measurement if premature ending)
  Difference = M6 -D0
  Variation % = 100 x (M6 - D0)/D0
HAD (Hospital Anxiety and Depression) scale | 6 months (or last measurement if premature ending)
  Qualitative analysis:
  * improvement from sub-score > 10 to sub-score < 10
  * no change
  * worsening from sub-score < 10 to sub-score > 10
Bladder diary | 6 Months (or last visit if premature ending)
  A bladder diary will be filled by the patient for 3 days before the inclusion visit and then for 3 days before the final visit.
  The following items will be compared between D0 and M6: normal urinary episodes, incontinence episodes and drinks, in number and volume.
  Difference = M6 - D0 Variation % = 100 x (M6-D0)/D0

OTHER OUTCOMES:
Adverse Events | 6 Months
Compliance | 6 Months
  The lasts electro-stimulation sessions are recorded by the medical device.

CONTACTS AND LOCATIONS:
Overall Officials: Marc Bernardini, MD, Principal Investigator
Locations (1):
- Marc Bernardini, Marseille, France